CLINICAL TRIAL: NCT03940144
Title: Department of Anesthesiology, Beijing Tong Ren Hospital Capital Medical University
Brief Title: Effect of SVV-guided Fluid Therapy on Outcomes After Major Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, YANXIA SUN, staff anesthesiologist, Beijing Tongren Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PX2018007
Record Dates: First submitted 2019-04-25; First posted 2019-05-07 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Goal-directed Fluid Therapy

STUDY DESIGN:
Intervention Model Description: goal-directed fluid therapy guided by stroke volume variation and cardiac index using FloTrac/Vigileo monitor
Who Masked: Participant, Outcomes Assessor
Masking Description: Care providers and investigators in the operating room could not be blinded due to the presence of the cardiac index trending monitor. The postoperative assessors were blinded to the allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- goal-directed fluid therapy (Experimental): Stroke Volume variation (SVV)-guided fluid therapy
  Interventions: Device: the enhanced flow-based hemodynamic parameters of the FloTrac/Vigileo device
- Conventional fluid therapy (Active Comparator): Conventional fluid therapy such as CVP and MAP guided fluid therapy
  Interventions: Device: the enhanced flow-based hemodynamic parameters of the FloTrac/Vigileo device

INTERVENTIONS:
Device: the enhanced flow-based hemodynamic parameters of the FloTrac/Vigileo device — Stroke volume variation (SVV)-guided fluid therapy

SUMMARY:
The investigators conduct this randomized assessor-blinded controlled trial to evaluate the effect of SVV-guided fluid therapy on postoperative morbidity and mortality in comparison with conventional fluid therapy after major abdominal surgery. Half of participants will receive GDFT perioperatively, and the others will receive conventional fluid therapy

DETAILED DESCRIPTION:
Perioperative fluid management has been recognized as an important factor with an impact on postoperative recovery following major abdominal surgery. However, the optimal fluid management is difficult to achieve using standard parameters (e.g., heart rate [HR], blood pressure [BP], central venous pressure[CVP], or urine output) that poorly estimate preload and preload responsiveness. Goal-directed fluid therapy (GDFT) was proposed by introducing different hemodynamic variables into a dynamic perspective of individual fluid loading with or without vasoactive substances to reach predefined goal of optimal preload and/or oxygen delivery.There have been increasing numbers of studies evaluating the effect of perioperative GDFT on postoperative recovery following major abdominal surgery. However, the evidence for the beneficial effect of GDFT on postoperative recovery remains inconsistent.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (aged 18 to 80 years)
2. ASA I~III
3. BMI:18~30kg／m2
4. Procedures were considered major if listed for resection of gastrointestinal, gynecologic, and urologic cancer with tumor debulking, staging or reconstruction with a risk for significant surgical blood loss

Exclusion Criteria:

1. Patients under 18 years,
2. pregnant or lactating woman
3. patients with esophageal or gastric surgical history
4. co-existing congestive heart failure; chronic lung disease; or renal or hepatic dysfunction (creatinine >50 % or liver enzymes >50 % of normal values), and arrhythmias-operative down staging using chemotherapy and/or radiation therapy
5. patients undergoing emergency surgery
6. patients with co-existing congestive heart failure; chronic lung disease; or renal or hepatic dysfunction (creatinine >50 % or liver enzymes >50 % of normal values), and arrhythmias

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | from the end of surgery to discharge from hospital up to 30 days after surgery
  from the end of surgery to discharge from hospital
GI function | from the end of surgery to 30 days after surgery
  number of participants with I-FEED score >6

SECONDARY OUTCOMES:
mortality | from the end of surgery to 1 year after surgery
  death after surgery
postoperative pain score | 1 day, 3 days and 5 days after surgery
  VAS for pain :0 no pain and 10 for worst pain
postoperative recovery quality | 1 day, 3 days and 5 days after surgery
  QoR-15 :quality of recovery score : 0 worst recovery quality and 150 for best recovery
Postoperative complications | from end of surgery to 30 days after surgery
  number of any complications after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yanxia Sun, M.D., Principal Investigator — Beijing Tong Ren Hospital
Locations (1):
- Beijing Tongren Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sun Y, Liang X, Chai F, Shi D, Wang Y. Goal-directed fluid therapy using stroke volume variation on length of stay and postoperative gastrointestinal function after major abdominal surgery-a randomized controlled trial. BMC Anesthesiol. 2023 Dec 4;23(1):397. doi: 10.1186/s12871-023-02360-1. PMID 38049713